CLINICAL TRIAL: NCT03337984
Title: Damage Control Surgery in the Treatment of Hinchey Stage III and IV Diverticulitis: an Italian Nationwide Survey
Brief Title: Damage Control Surgery in the Treatment of Complicated Diverticulitis
Acronym: DACSCOD
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianluca Costa, Study Creator and Director, University of Roma La Sapienza
Other Study IDs: EM-SURG AOSA 2017_1
Record Dates: First submitted 2017-06-12; First posted 2017-11-09 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Diverticulitis
Keywords: Diverticulitis; Damage Control Surgery
MeSH Terms: conditions — Diverticulitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the use of damage control surgery by performing bowel resection and laparostomy in the treatment of Hinchey III or IV diverticulitis.

DETAILED DESCRIPTION:
Despite the progress in the resuscitation modalities of septic patients, Hartmann procedure (HP) is still considered the safest treatment for generalized peritonitis as a consequence of a complicated acute diverticulitis (stages III and IV of the Hinchey's classification). Almost the half of those patients do not have their stoma reversed because of its association with significant morbidity and mortality. To date, the use of resection with primary anastomosis (PA) is a matter of debate, as it is reported in the literature that it is substantially equivalent to HP in terms of morbidity and length of postoperative stay. For these reason, PA is often reserved for younger patients with few co-morbidities and a lesser degree of peritoneal contamination. In the last decade, Damage Control Surgery has been emerging as a valid alternative to HP and RA in patients presenting a severe sepsis caused by purulent or fecal peritonitis in acute diverticulitis. Initially described for the treatment of major abdominal injuries, indications for DCS have subsequently been extended to septic shock, abdominal compartment syndrome and impossibility to perform a primary closure. However, there is still no consensus about the use of DCS in perforated acute diverticulitis.

The aim of this study was to describe "how-to-use" the Damage Control Surgery in patients with purulent and fecal peritonitis following a severe acute diverticulitis and report the impact on patients' outcomes after the application of this technique in several Italian centers of emergency surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for Hinchey III and IV stage scheduled for immediate Hartmann's procedure and ICU recovery

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated on for Hinchey III or IV class and treated by damage control surgery procedure
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Mortality | 6 months
  Mortality rate related to treatment

SECONDARY OUTCOMES:
Morbidity | 6 months
  Complications rate arranged by Clavien-Dindo classification I to IV
Lenght of stay (LOS) | 6 months
  Days of stay as inpatient
ICU lenght of stay | 12 months
  Days of stay as
Number of Hartmann's procedure | 1 month
  Observed to expected (O:E) ratio of Hartmann's procedures

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Costa, MD, PhD, Study Director — University of Roma La Sapienza, Sant' Andrea University Hospital
Locations (9):
- Italy (9):
  - Policlinico San Pietro, Ponte San Pietro, Bergamo
  - Azienda Ospedaliera Cardarelli, Napoli, Campania
  - Ospedale Civile di Adria, Adria, Rovigo
  - Azienda Ospedaliero Universitaria Ospedale Riuniti Ancona, Ancona, The Marches
  - Ospedale San Donato, Arezzo, Tuscany
  - Azienda Ospedaliera Pisana Policlinico Universitario Cisanello, Pisa, Tuscany
  - Ospedale San Giovanni Battista, Foligno, Umbria
  - Azienda Ospedaliera Santa Maria, Terni, Umbria
  - Policlinico Abano Terme, Abano Terme, Veneto

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will probably be shared with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Since six months from study start to six months from study completion
Access Criteria: By request

REFERENCES:
- [Background] Costa G, La Torre M, Frezza B, Fransvea P, Tomassini F, Ziparo V, Balducci G. Changes in the surgical approach to colonic emergencies during a 15-year period. Dig Surg. 2014;31(3):197-203. doi: 10.1159/000365254. Epub 2014 Aug 28. PMID 25170867
- [Background] Ince M, Stocchi L, Khomvilai S, Kwon DS, Hammel JP, Kiran RP. Morbidity and mortality of the Hartmann procedure for diverticular disease over 18 years in a single institution. Colorectal Dis. 2012 Aug;14(8):e492-8. doi: 10.1111/j.1463-1318.2012.03004.x. PMID 22356208
- [Background] Turley RS, Barbas AS, Lidsky ME, Mantyh CR, Migaly J, Scarborough JE. Laparoscopic versus open Hartmann procedure for the emergency treatment of diverticulitis: a propensity-matched analysis. Dis Colon Rectum. 2013 Jan;56(1):72-82. doi: 10.1097/DCR.0b013e3182749cf5. PMID 23222283
- [Background] Benz D, Balogh ZJ. Damage control surgery: current state and future directions. Curr Opin Crit Care. 2017 Dec;23(6):491-497. doi: 10.1097/MCC.0000000000000465. PMID 29035926
- [Background] Girard E, Abba J, Boussat B, Trilling B, Mancini A, Bouzat P, Letoublon C, Chirica M, Arvieux C. Damage Control Surgery for Non-traumatic Abdominal Emergencies. World J Surg. 2018 Apr;42(4):965-973. doi: 10.1007/s00268-017-4262-6. PMID 28948335
- [Background] Bruns BR, Ahmad SA, O'Meara L, Tesoriero R, Lauerman M, Klyushnenkova E, Kozar R, Scalea TM, Diaz JJ. Nontrauma open abdomens: A prospective observational study. J Trauma Acute Care Surg. 2016 Apr;80(4):631-6. doi: 10.1097/TA.0000000000000958. PMID 26808023
- [Background] Weber DG, Bendinelli C, Balogh ZJ. Damage control surgery for abdominal emergencies. Br J Surg. 2014 Jan;101(1):e109-18. doi: 10.1002/bjs.9360. Epub 2013 Nov 25. PMID 24273018
- [Background] Khan A, Hsee L, Mathur S, Civil I. Damage-control laparotomy in nontrauma patients: review of indications and outcomes. J Trauma Acute Care Surg. 2013 Sep;75(3):365-8. doi: 10.1097/TA.0b013e31829cb65e. PMID 23928745
- [Background] Subramanian A, Balentine C, Palacio CH, Sansgiry S, Berger DH, Awad SS. Outcomes of damage-control celiotomy in elderly nontrauma patients with intra-abdominal catastrophes. Am J Surg. 2010 Dec;200(6):783-8; discussion 788-9. doi: 10.1016/j.amjsurg.2010.07.027. PMID 21146021
- [Background] Cirocchi R, Arezzo A, Vettoretto N, Cavaliere D, Farinella E, Renzi C, Cannata G, Desiderio J, Farinacci F, Barberini F, Trastulli S, Parisi A, Fingerhut A. Role of damage control surgery in the treatment of Hinchey III and IV sigmoid diverticulitis: a tailored strategy. Medicine (Baltimore). 2014 Nov;93(25):e184. doi: 10.1097/MD.0000000000000184. PMID 25437034
- [Background] Cassini D, Miccini M, Manoochehri F, Gregori M, Baldazzi G. Emergency Hartmann's Procedure and Its Reversal: A Totally Laparoscopic 2-Step Surgery for the Treatment of Hinchey III and IV Diverticulitis. Surg Innov. 2017 Dec;24(6):557-565. doi: 10.1177/1553350617722226. Epub 2017 Jul 27. PMID 28748737
- [Background] Bridoux V, Regimbeau JM, Ouaissi M, Mathonnet M, Mauvais F, Houivet E, Schwarz L, Mege D, Sielezneff I, Sabbagh C, Tuech JJ. Hartmann's Procedure or Primary Anastomosis for Generalized Peritonitis due to Perforated Diverticulitis: A Prospective Multicenter Randomized Trial (DIVERTI). J Am Coll Surg. 2017 Dec;225(6):798-805. doi: 10.1016/j.jamcollsurg.2017.09.004. Epub 2017 Sep 22. PMID 28943323
- [Background] Coccolini F, Montori G, Ceresoli M, Catena F, Moore EE, Ivatury R, Biffl W, Peitzman A, Coimbra R, Rizoli S, Kluger Y, Abu-Zidan FM, Sartelli M, De Moya M, Velmahos G, Fraga GP, Pereira BM, Leppaniemi A, Boermeester MA, Kirkpatrick AW, Maier R, Bala M, Sakakushev B, Khokha V, Malbrain M, Agnoletti V, Martin-Loeches I, Sugrue M, Di Saverio S, Griffiths E, Soreide K, Mazuski JE, May AK, Montravers P, Melotti RM, Pisano M, Salvetti F, Marchesi G, Valetti TM, Scalea T, Chiara O, Kashuk JL, Ansaloni L. The role of open abdomen in non-trauma patient: WSES Consensus Paper. World J Emerg Surg. 2017 Aug 14;12:39. doi: 10.1186/s13017-017-0146-1. eCollection 2017. PMID 28814969
- [Background] Kafka-Ritsch R, Birkfellner F, Perathoner A, Raab H, Nehoda H, Pratschke J, Zitt M. Damage control surgery with abdominal vacuum and delayed bowel reconstruction in patients with perforated diverticulitis Hinchey III/IV. J Gastrointest Surg. 2012 Oct;16(10):1915-22. doi: 10.1007/s11605-012-1977-4. Epub 2012 Jul 28. PMID 22843083
- [Background] Perathoner A, Klaus A, Muhlmann G, Oberwalder M, Margreiter R, Kafka-Ritsch R. Damage control with abdominal vacuum therapy (VAC) to manage perforated diverticulitis with advanced generalized peritonitis--a proof of concept. Int J Colorectal Dis. 2010 Jun;25(6):767-74. doi: 10.1007/s00384-010-0887-8. Epub 2010 Feb 11. PMID 20148255
- [Background] Sohn M, Agha A, Heitland W, Gundling F, Steiner P, Iesalnieks I. Damage control strategy for the treatment of perforated diverticulitis with generalized peritonitis. Tech Coloproctol. 2016 Aug;20(8):577-83. doi: 10.1007/s10151-016-1506-7. Epub 2016 Jul 22. PMID 27448296
- [Background] Hess GF, Schafer J, Rosenthal R, Kettelhack C, Oertli D. Reversal after Hartmann's procedure in patients with complicated sigmoid diverticulitis. Colorectal Dis. 2017 Jun;19(6):582-588. doi: 10.1111/codi.13553. PMID 27805772
- [Background] Vennix S, Boersema GS, Buskens CJ, Menon AG, Tanis PJ, Lange JF, Bemelman WA. Emergency Laparoscopic Sigmoidectomy for Perforated Diverticulitis with Generalised Peritonitis: A Systematic Review. Dig Surg. 2016;33(1):1-7. doi: 10.1159/000441150. Epub 2015 Nov 10. PMID 26551040
- [Background] Richards CH, Roxburgh CS; Scottish Surgical Research Group (SSRG). Surgical outcome in patients undergoing reversal of Hartmann's procedures: a multicentre study. Colorectal Dis. 2015 Mar;17(3):242-9. doi: 10.1111/codi.12807. PMID 25331720
- [Background] Horesh N, Lessing Y, Rudnicki Y, Kent I, Kammar H, Ben-Yaacov A, Dreznik Y, Tulchinsky H, Avital S, Mavor E, Wasserberg N, Kashtan H, Klausner JM, Gutman M, Zmora O. Considerations for Hartmann's reversal and Hartmann's reversal outcomes-a multicenter study. Int J Colorectal Dis. 2017 Nov;32(11):1577-1582. doi: 10.1007/s00384-017-2897-2. Epub 2017 Sep 6. PMID 28879552